CLINICAL TRIAL: NCT03694535
Title: Intravesical Mitomycin-C With Bladder Wall Hyperthermia in Intermediate and High Risk Non-muscle Invasive Bladder Cancer
Brief Title: Intravesical Thermochemotherapy With Mitomycin-c
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Abdullah Demirtas, Md, Assoc. Prof., TC Erciyes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014/387
Record Dates: First submitted 2018-09-27; First posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Bladder Cancer
Keywords: Thermochemotherapy; bladder; cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Intervention Model Description: single group of patients composed of intermediate and high risk non muscle invasive bladder cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bladder wall thermochemotherapy (Experimental): Mitomycin-C application with bladder wall thermochemotherapy system after TUR bladder tumor in intermediate and high risk non muscle invasive bladder cancer
  Interventions: Drug: bladder wall thermotherapy with Mitomycin-c

INTERVENTIONS:
Drug: bladder wall thermotherapy with Mitomycin-c — application of intravesical mitomycin-C with hyperthermia

SUMMARY:
To investigate effect of intravesical mitomycin-C(MMC) applied with bladder wall thermotherapy system on reccurrence and progression status of intermediate and high risk non muscle invasive bladder cancer

DETAILED DESCRIPTION:
Before the application of TCT, complete transurethral bladder tumour resection (TURBT) was performed. RE-TURBT was conducted within 4 weeks for patients with initial T1 pathology. The first TCT instillation was applied at 1mo following the TURBT or the RE-TURBT.

Thermochemotherapy application and treatment schedule:

The bladder wall TCT (BWT) system (Elmedical Ltd, Hod-Hasharon, Israel) was used as a conductive heating modality. MMC (40 mg; MMC Kyowa Hakko Kogyo Co., Ltd., Tokyo, Japan) was mixed with 50 mL of 0.9% saline solution and applied using a disposable silicone 20Fr 3-way TCT catheter (UniThermia catheter; Elmedical Ltd). In each session, the bladder was irrigated with MMC solution at 42°C-45°C for 45 min via the BWT system. The treatment schedule consisted of an initial 6-week instillation, followed by control cystoscopy and urine cytology in the 3rd month and monthly instillations up to 1 yr. Urine cytology and cystoscopy were performed every three months. The samples were collected from the suspected areas during cystoscopy. At the end of the first year, control cystoscopy with random bladder biopsies was conducted. During the second year, routine controls were conducted every three months. Subsequently, follow-ups were performed every six months. In case of development of any complication in a patient, TCT was discontinued. Before each instillation of TCT, clear urine cultures were obtained from all patients. No prophylactic anticholinergic was administered prior to intravesical TCT. If TUR BT pathology was Ta or T1 during the follow-up, it was accepted as a recurrence. If it was CIS or T2, it was accepted as a progression. All adverse events observed during the study were recorded according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 [9. All study protocols were approved by the local ethical committee at our institution. An informed consent was obtained from all patients.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed or followed as recurrent intermediate-risk non muscle invasive non muscle invasive bladder cancer according to the criteria of European Association of Urology.
* newly diagnosed or followed as recurrent high-risk non muscle invasive non muscle invasive bladder cancer according to the criteria of European Association of Urology.
* pathology of urothelial carcinoma

Exclusion Criteria:

* Low bladder capacity (<150ml)
* increased post voiding residual urine (>150ml)
* untreatable or uncontrollable urinary tract infection
* history of urethral stricture
* presence of bladder diverticula larger than 1 cm
* pathology other than urothelial carcinoma
* WHO (World Health Organization) performance status > 2
* upper urinary tract urothelial carcinoma diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Recurrence | From the beginning of thermochemoterapy until the date of first documented recurrence assessed up to 2 years
  recurrence rate of non muscle invasive bladder cancer during or after treatment
Progression rate | From the beginning of thermochemoterapy until the date of first documented progression assessed up to 2 years
  progression rate of non muscle invasive bladder cancer during or after treatment ( progress to muscle invasive stage or carcinoma in situ)

SECONDARY OUTCOMES:
Side effects | From the beginning of thermochemoterapy until the date of first documented side effect(s) assessed up to 2 years
  side effects detected during TCT instillation

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Demirtas, MD, Principal Investigator — TC Erciyes University Medical Faculty
Locations (1):
- Department of Urology, Ercieys University, Faculty Of Medicine,, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moskovitz B, Meyer G, Kravtzov A, Gross M, Kastin A, Biton K, Nativ O. Thermo-chemotherapy for intermediate or high-risk recurrent superficial bladder cancer patients. Ann Oncol. 2005 Apr;16(4):585-9. doi: 10.1093/annonc/mdi124. Epub 2005 Feb 25. PMID 15734775
- [Background] Colombo R, Salonia A, Leib Z, Pavone-Macaluso M, Engelstein D. Long-term outcomes of a randomized controlled trial comparing thermochemotherapy with mitomycin-C alone as adjuvant treatment for non-muscle-invasive bladder cancer (NMIBC). BJU Int. 2011 Mar;107(6):912-8. doi: 10.1111/j.1464-410X.2010.09654.x. Epub 2010 Oct 4. PMID 21029314